CLINICAL TRIAL: NCT04619641
Title: Physiological Effects of a New Interface Combining High-flow Nasal Cannula and Cpap on Lung Ventilation and Gas Distribution in Patients With Mild-to-moderate Acute Respiratory Distress Syndrome: a Pilot Study
Brief Title: Physiological Effects of a New Interface on Lung Ventilation and Gas Distribution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Prof, University Magna Graecia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OptiPAP EIT
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High flow nasal cannula (HFNC) (Active Comparator): HFNC will be applied by means of a dedicated device (AIRVO2, Fisher & Paykel Healthcare, Auckland, New Zealand). Gas flow will be set at 50 L/min, and humidification chamber will be set at 31°C.
  Interventions: Device: High Flow Nasal Cannula (HFNC)
- Continuous Positive Airway Pressure (CPAP) (Active Comparator): CPAP will be delivered through a helmet (Castar Next, Intersurgical S.p.A., Mirandola, Italy), with an adjustable Positive End-Expiratory Pressure (PEEP) valve (2.5-20 cmH2O) set at 10 cmH2O (Intersurgical S.p.A., Mirandola, Italy). The helmet will be connected to a turbine-driven ventilator (Monnal T60, Air Liquide Medical Systems, Antony, France) set to deliver oxygen-air admixture at a continuous flow rate of 60 L/min, in order to improve CO2 wash out. No heated humidification will be applied to avoid the "fog effect" in the helmet.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- HFNC+CPAP (Active Comparator): HFNC+CPAP consists in the contemporaneous application of HFNC and CPAP through helmet. HFNC will be set at 30 L/min, with a temperature at 31° C and 100% of relative humidity, while CPAP will be delivered through a helmet (Castar Next, Intersurgical S.p.A., Mirandola, Italy), with an adjustable Positive End-Expiratory Pressure (PEEP) valve (2.5-20 cmH2O) set at 10 cmH2O (Intersurgical S.p.A., Mirandola, Italy). The helmet will be connected to a turbine-driven ventilator (Monnal T60, Air Liquide Medical Systems, Antony, France) set to deliver oxygen-air admixture at a continuous flow rate of 60 L/min, in order to improve CO2 wash out. No heated humidification will be applied to avoid the "fog effect" in the helmet
  Interventions: Device: High Flow Nasal Cannula (HFNC); Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: High Flow Nasal Cannula (HFNC) — HFNC will be set at 30 L/min, with a temperature at 31° C and 100% of relative humidity
  Arms: HFNC+CPAP; High flow nasal cannula (HFNC)
Device: Continuous Positive Airway Pressure (CPAP) — CPAP will be delivered through a helmet (Castar Next, Intersurgical S.p.A., Mirandola, Italy), with an adjustable Positive End-Expiratory Pressure (PEEP) valve (2.5-20 cmH2O) set at 10 cmH2O (Intersurgical S.p.A., Mirandola, Italy). The helmet will be connected to a turbine-driven ventilator (Monnal T60, Air Liquide Medical Systems, Antony, France) set to deliver oxygen-air admixture at a continuous flow rate of 60 L/min, in order to improve CO2 wash out. No heated humidification will be applied to avoid the "fog effect" in the helmet
  Arms: Continuous Positive Airway Pressure (CPAP); HFNC+CPAP

SUMMARY:
Hypoxemic Acute Respiratory Failure (hARF) is a common reason of admission to Intensive Care. Different modalities can be used to administer oxygen, which is the first supportive treatment in these patients. Recently a new device combining high flow nasal cannula (HFNC) and continuous positive airway pressure (CPAP) has been developed, but a few is known in these patients.

Investigators have designed this pilot physiologic randomized cross-over study to assess, in patients with hARF, the effects of a new device combining high-flow oxygen through nasal cannula (HFNC) and continuous positive airway pressure (CPAP) on lung aeration and ventilation distribution .

DETAILED DESCRIPTION:
Around 30% of patients admitted to the Intensive Care Unit (ICU) are affected by hypoxemic Acute Respiratory Failure (hARF). The primary supportive treatment in hypoxemic patients is oxygen therapy, which is commonly delivered through nasal prongs or masks. New devices, able to deliver high-flow gas through a nasal cannula (HFNC), have been recently made available. HFNC delivers heated and humidified gas up to 60 L/min, with a fraction of inspired oxygen (FiO2) ranging from 0.21 to 1, via a wide bore soft nasal prong. Warming and humidification of the inspired gas prevent the adverse effects of cool dry gases on the airway epithelium and facilitate expectoration. HFNC also washes out exhaled carbon dioxide (CO2) from the pharyngeal dead space. HFNC has been shown an effective means to deliver oxygen therapy in many clinical conditions.

In healthy subject during spontaneous unassisted breathing, end-expiratory pharyngeal pressure is about 0.3 and 0.8 cmH2O, with open and closed mouth, respectively. Compared to unassisted spontaneous breathing, HFNC generates greater pharyngeal pressure during expiration, while in the course of inspiration it drops to zero, which limits the effectiveness of HFNC in patients with lung edema and/or collapse. By recruiting lung atelectatic regions, reducing venous admixture and decreasing the inspiratory effort, continuous positive airway pressure (CPAP) is likely more effective in these instances. Compared to noninvasive ventilation by application of an inspiratory pressure support, CPAP offers several advantages, which include ease of use and lack of patient-ventilator asynchrony.

CPAP may be applied either through mask or helmet. This latter is better tolerated than facial masks and allows more prolonged continuous CPAP application. When applying CPAP by helmet, however, heating and humidification of the inhaled gas is problematic because of condensation of water inside the interface, so called "fog effect". Moreover, in patients receiving CPAP by helmet some re-breathing occurs.

To overcome these limitations and combine the beneficial effects of HFNC and CPAP, investigators designed a new device combining HFNC and helmet CPAP.

Recently, it has been found this combination capable to provide a stable CPAP and effective CO2 washout from the upper airways with negligible CO2 re-breathing. Nonetheless, because of the complex interplay between CPAP and HFNC, the amount of truly applied airway pressure, diaphragm function and temperature inside the helmet might be affected to some extent. In 14 adult healthy volunteers, we found that adding HFNC to CPAP (as referenced to CPAP), 1) did not importantly alter either the pre-set airway pressure during inspiration or temperature inside the helmet; 2) increased expiratory airway pressure proportionally to the flow administered by HFNC, but to a lower extent than HFNC alone (as referenced to spontaneous breathing); 3) determined only slight modifications of the respiratory drive (as assessed through diaphragm ultrasound), compared to CPAP alone, 4) did not cause "fog effect" inside the helmet and 5) did not worsen comfort. We therefore suggested that adding heated humidified air through nasal cannula at a flow of 30 L/min during CPAP would probably be the best setting to be applied in patients with hypoxemic acute respiratory failure.

Electrical Impedance Tomography (EIT) is a non-invasive bedside monitoring device aimed at assessing lung aeration and ventilation. HFNC and CPAP devices was shown to modify lung aeration and ventilation in patients with hARF. However, nothing is known about the effect of the combination of HFNC+CPAP on lung ventilation in patients with hARF. Investigators have therefore designed this pilot physiologic randomized cross-over study to investigate the effects of HFNC+CPAP on lung aeration and ventilation distribution, gas exchange and patient's comfort.

ELIGIBILITY:
Inclusion Criteria:

* presence of hypoxemic Acute Respiratory Failure
* absence of history of chronic respiratory failure or moderate-to-severe cardiac insufficiency

Exclusion Criteria:

* reduced level of consciousness, as indicated by a Glasgow Coma Scale < 12
* severe respiratory distress (i.e. respiratory rate > 35 breaths/min)
* hemodynamic instability, (i.e. systolic arterial pressure <90 mmHg or mean systolic pressure <65 mmHg despite fluid repletion)
* need for vasoactive agents, i.e. vasopressin or epinephrine at any dosage, or norepinephrine >0.3 mcg/kg/min or dobutamine>5 mcg/kg/min
* life-threatening arrhythmias or electrocardiographic signs of ischemia
* acute respiratory failure secondary to neurological disorders, status asthmaticus, chronic obstructive pulmonary disease (COPD), cardiogenic pulmonary oedema
* presence of tracheotomy
* uncontrolled vomiting
* more than 2 acute organ failures
* body mass index >30 kg/m2
* documented history or suspicion of obstructive sleep apnoea
* facial anatomy contraindicating helmet or nasal cannula application
* contraindications to placement of EIT (i.e., pneumothorax, pulmonary emphysema, chest burns or thoracic surgery within 1 week)
* inclusion in other research protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of end-expiratory lung impedance (dEELI) from HFNC | After 30 minutes of treatment application
  change from HFNC, expressed in percentage of the tidal volume, of the end expiratory lung volume as assessed through electrical impedance tomography

SECONDARY OUTCOMES:
Global Inhomogeneity (GI) | After 30 minutes of treatment application
  inhomogeneity of air distribution within the lung as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from HFNC | After 30 minutes of treatment application
  change from HFNC, expressed in percentage, of the tidal volume as assessed through electrical impedance tomography
Arterial partial pressure of oxygen (PaO2) | After 30 minutes of treatment application
  Analysis of arterial blood gases
Arterial partial pressure of carbon dioxide (PaCO2) | After 30 minutes of treatment application
  Analysis of arterial blood gases
Patient's comfort | After 30 minutes of treatment application
  It will be measured using an 11-point Numeric Rating Scale. Briefly, after detailed explanation before initiating the protocol, patients will be asked to indicate a number between 0 (worst possible comfort) and 10 (no discomfort) on an adapted printed scale.
Patient's Dyspnea | After 30 minutes of treatment application
  It will be measured using an 11-point Numeric Rating Scale. Briefly, after detailed explanation before initiating the protocol, patients will be asked to indicate a number between 0 (no dyspnoea) and 10 (worst possible dyspnoea) on an adapted printed scale.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University, Anesthesia and Intensive Care Unit

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data will be anonymously shared after reasonable request to the Principal Investigator or Corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study and results publication on an international medical journal
Access Criteria: On reasonable request to the corresponding author or principal investigator

REFERENCES:
- [Background] Garofalo E, Bruni A, Pelaia C, Cammarota G, Murabito P, Biamonte E, Abdalla K, Longhini F, Navalesi P. Evaluation of a New Interface Combining High-Flow Nasal Cannula and CPAP. Respir Care. 2019 Oct;64(10):1231-1239. doi: 10.4187/respcare.06871. Epub 2019 Jun 4. PMID 31164484
- [Background] Mauri T, Spinelli E, Mariani M, Guzzardella A, Del Prete C, Carlesso E, Tortolani D, Tagliabue P, Pesenti A, Grasselli G. Nasal High Flow Delivered within the Helmet: A New Noninvasive Respiratory Support. Am J Respir Crit Care Med. 2019 Jan 1;199(1):115-117. doi: 10.1164/rccm.201806-1124LE. No abstract available. PMID 30240275
- [Background] Grieco DL, Menga LS, Raggi V, Bongiovanni F, Anzellotti GM, Tanzarella ES, Bocci MG, Mercurio G, Dell'Anna AM, Eleuteri D, Bello G, Maviglia R, Conti G, Maggiore SM, Antonelli M. Physiological Comparison of High-Flow Nasal Cannula and Helmet Noninvasive Ventilation in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2020 Feb 1;201(3):303-312. doi: 10.1164/rccm.201904-0841OC. PMID 31687831